CLINICAL TRIAL: NCT01287936
Title: A Phase 1/2A Study of the Safety and Efficacy of Modified Stromal Cells (SB623) in Patients With Stable Ischemic Stroke
Brief Title: A Study of Modified Stem Cells in Stable Ischemic Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SanBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SB-STR01
Record Dates: First submitted 2011-01-27; First posted 2011-02-02 (Estimated); Results first posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Chronic Ischemic Stroke
Keywords: Chronic Stroke; Stable Stroke; Ischemic Stroke; Fixed Motor Deficits
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SB623 Implant (2.5M) (Experimental): 2.5 million SB623 cells
  Interventions: Biological: SB623
- SB623 Implant (5.0M) (Experimental): 5 million SB623 cells
  Interventions: Biological: SB623
- SB623 Implant (10.0M) (Experimental): 10 million SB623 cells
  Interventions: Biological: SB623

INTERVENTIONS:
Biological: SB623 — SB623, a modified stem-cell product

SUMMARY:
The primary purpose of the clinical study is to determine the safety of a modified stem cell SB623 when administered to chronic, stable ischemic stroke patients. A second purpose is to determine whether SB623 might improve stroke symptoms. Chronic, stable ischemic stroke patients must be between 6 and 60 months after their stroke, and with only this one prior stroke, and with no further improvement from physical therapy.

DETAILED DESCRIPTION:
Chronic, stable stroke patients have no existing alternative treatments after rehabilitation therapy. SB623, a modified stem cell preparation, has been shown to improve motor function when administered in animal models of stable stroke. Safety studies in animals have shown no adverse events attributed to SB623. Patients who meet the entry criteria for this study will have regular examinations, radiological evaluations (CT, MRI, PET), and be followed for two years. Regular neurological evaluations will also be done using standard questionnaires, with occasional video recording if improvements are evident. Key entry criteria for this study, in addition to 6-60 months post-ischemic stroke, include moderately severe symptoms--e.g., difficulty standing or walking, and/or difficulty using arms or hands, and/or speech impediments.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of one completed ischemic stroke in subcortical region of MCA or lenticulostriate artery with or without cortical involvement
* Between 6 and 60 months post-stroke, and having a motor neurological deficit
* No significant further improvement with physical therapy/rehabilitation
* Able and willing to undergo computed tomography (CT), magnetic resonance imaging (MRI), and positron-emission tomography (PET) scans of the head

Exclusion Criteria:

* History of more than 1 symptomatic stroke
* History of seizures
* History or presence of any other major neurological disease
* Myocardial infarction within prior 6 mos.
* Known presence of any malignancy except squamous or basal cell carcinoma of the skin
* Participation in any other investigational trial within 4 weeks of initial screening and within 7 weeks of study entry
* Contraindications to head CT, MRI, or PET
* Pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary K Steinberg, M.D., Ph.D., Principal Investigator — Stanford University; Lawrence R Wechsler, M.D., Principal Investigator — University of Pittsburgh Medical Center; Joshua M Rosenow, M.D.,FACS, Principal Investigator — Northwestern University Feinberg School of Medicine; James Markert, M.D., Principal Investigator — University of Alabama at Birmingham; Robert E Gross, M.D., Ph.D., Principal Investigator — Emory University
Locations (5):
- United States (5):
  - University of Alabama, Birmingham, Alabama
  - Stanford University School of Medicine, Stanford, California
  - Emory University, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Steinberg GK, Kondziolka D, Wechsler LR, Lunsford LD, Kim AS, Johnson JN, Bates D, Poggio G, Case C, McGrogan M, Yankee EW, Schwartz NE. Two-year safety and clinical outcomes in chronic ischemic stroke patients after implantation of modified bone marrow-derived mesenchymal stem cells (SB623): a phase 1/2a study. J Neurosurg. 2018 Nov 23;131(5):1462-1472. doi: 10.3171/2018.5.JNS173147. Print 2019 Nov 1. PMID 30497166
- [Derived] Steinberg GK, Kondziolka D, Wechsler LR, Lunsford LD, Coburn ML, Billigen JB, Kim AS, Johnson JN, Bates D, King B, Case C, McGrogan M, Yankee EW, Schwartz NE. Clinical Outcomes of Transplanted Modified Bone Marrow-Derived Mesenchymal Stem Cells in Stroke: A Phase 1/2a Study. Stroke. 2016 Jul;47(7):1817-24. doi: 10.1161/STROKEAHA.116.012995. Epub 2016 Jun 2. PMID 27256670

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | SB623 Implant (10.0M)
Started | 6 | 6 | 6
Completed | 6 | 5 | 5
Not Completed | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | SB623 Implant (10.0M) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (7.62) | 67.2 (7.60) | 56.8 (13.30) | 61.3 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 3 | 2 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 3 | 4 | 5 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs)
Description: Number of subjects with TEAEs by maximum severity. The severity of all AEs was assessed by the Investigator using the World Health Organization (WHO) Toxicity Scale. For abnormalities not found elsewhere in the WHO table, the following scale was used to assign severity:
  Mild: Transient mild discomfort; no limitation in activity; no medical intervention/therapy required.
  Moderate: Mild-to-moderate limitation in activity; some assistance may be need. No or minimal medical intervention/therapy required.
  Severe: Marked limitation in activity, some assistance usually required; medical intervention/therapy required; hospitalization or prolongation of current hospitalization possible.
  Life-threatening: Extreme limitation in activity, significant assistance required; significant medial intervention/therapy required; hospitalization or prolongation of current hospitalization or hospice care probable.
Time Frame: 6 months
Population: Safety population includes all enrolled patients who have received study treatment and who have any post-baseline data.
Measure: Count of Participants; unit: Participants
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | SB623 Implant (10.0M)
Number analyzed (Participants) | 6 | 6 | 6
Participants
  Mild | 1 | 1 | 0
  Moderate | 3 | 2 | 4
  Severe | 1 | 3 | 2
  Life threatening | 1 | 0 | 0

2. Secondary Outcome: Change in the European Stroke Scale (ESS) Total Score From Baseline at Month 6
Description: The ESS is the sum of 14 items that are used to assess a patient who has recently had a stroke. These 14 items are level of consciousness, comprehension, speech, visual field, gaze, facial movement, arm in outstretched position, arm raising, extension of the wrist, fingers, leg maintained in position, leg flexing, dorsiflexion of the foot, and gait. A certain number of points are given for each parameter. The range of the total score of ESS is 0 - 100, with a completely normal person having a score of 100 and maximally affected person with a score of zero.
Time Frame: 6 months
Population: Intent-to-Treat (ITT) Population: Included all randomized subjects who completed the surgery treatment procedure (18 subjects).
Measure: Mean (Standard Deviation); unit: Change in score on a scale from baseline
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | SB623 Implant (10.0M)
Number analyzed (Participants) | 6 | 6 | 6
Change in score on a scale from baseline | 7.67 (8.140) | 4.50 (5.244) | 7.75 (10.012)
Statistical Analysis 1: Comparison: SB623 Implant (2.5M) vs SB623 Implant (5.0M) vs SB623 Implant (10.0M); Test type: Superiority; p < 0.001, Wilcoxon Signed Rank test

3. Secondary Outcome: Change in the European Stroke Scale (ESS) Motor Function Total Score From Baseline at Month 6
Description: The ESS motor function score is a sum of the selected items: facial movement, arm in outstretched position, arm raising, extension of wrist, fingers, leg maintained in position, leg flexing, dorsiflexion of foot, and gait. A completely normal person will have a score of 66. The maximally affected person will have a score of zero.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in score on a scale from baseline
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | SB623 Implant (10.0M)
Number analyzed (Participants) | 6 | 6 | 6
Change in score on a scale from baseline | 6.33 (6.186) | 3.67 (3.933) | 6.25 (5.560)

4. Secondary Outcome: Change in the National Institutes of Health Stroke Scale (NIHSS) Total Score From Baseline at Month 6
Description: The NIHSS is a standardized method used to measure the level of impairment caused by a stroke. The scale consists of 11 items that measure several aspects of brain function, including consciousness, vision, sensation, movement, speech, and language. A certain number of points are given for each impairment uncovered during a focused neurological examination. A maximal score of 42 represents the most severe and devastating stroke with 0=no stroke, 1-4=minor stroke, 5-15=moderate stroke, 15-20=moderate/severe stroke, and 21-42=severe stroke.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: change in score on a scale from baseline
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | SB623 Implant (10.0M)
Number analyzed (Participants) | 6 | 6 | 6
change in score on a scale from baseline | -2.00 (1.265) | -0.83 (1.472) | -2.50 (3.512)
Statistical Analysis 1: Comparison: SB623 Implant (2.5M) vs SB623 Implant (5.0M) vs SB623 Implant (10.0M); Test type: Superiority; p = 0.004, Wilcoxon Signed Rank test

5. Secondary Outcome: Change in the National Institutes of Health Stroke Scale (NIHSS) Motor Function Total Score From Baseline at Month 6
Description: The NIHSS is a standardized method used to measure the level of impairment caused by a stroke. The NIHSS Motor Function Total Score consists of 3 items: motor arm, motor leg, and limb ataxia, with 0 = no stroke and a maximal score of 18 = most severe impairment for motor function.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: change in score on a scale from baseline
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | SB623 Implant (10.0M)
Number analyzed (Participants) | 6 | 6 | 6
change in score on a scale from baseline | -1.33 (0.816) | -0.83 (1.472) | -1.00 (1.414)

6. Secondary Outcome: Change in the Modified Rankin Scale (mRS) Response From Baseline at Month 6
Description: The mRS is a commonly used scale for measuring the degree of disability in daily activities for patients who have suffered a stroke. The mRS is an ordinal scale from 0 (no symptoms at all) to 5 (severe disability; requiring constant nursing care and attention, bedridden, incontinent) with a sixth category of death.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in score on a scale from baseline
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | SB623 Implant (10.0M)
Number analyzed (Participants) | 6 | 6 | 6
Change in score on a scale from baseline | 0 (0) | -0.17 (0.408) | -0.25 (0.500)

7. Secondary Outcome: Change in the Fugl-Meyer Total Score From Baseline at Month 6
Description: The Fugl-Meyer Scale is a stroke-specific, performance-based impairment index. The scale is comprised of 5 domains (motor score, sensation, balance, joint range of motion, and joint pain) with 155 items in total. Scoring is based on direct observation of performance. Scale items in all 5 domains are scored on the basis of ability to complete the item using a 3-point Likert-type ordinal scale, where 0=cannot perform, 1=performs partially, and 2=performs fully. Points are divided among the domains: (a) Motor performance [0 (hemiplegia) - 100 (normal motor performance) points]; (b) Balance [0-14 points: 6 for sitting; 8 for standing]; (c) Sensation [0-24 points: 8 for light touch; 16 for position sense]; (d) Joint range of motion [0-44 points]; (e) Joint pain [0-44 points]. For all domains, a maximally affected person will score 0 while a fully functional person will have the highest score. All items are summed to provide a minimum score of 0 and a maximum score of 226.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in score on a scale from baseline
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | SB623 Implant (10.0M)
Number analyzed (Participants) | 6 | 6 | 6
Change in score on a scale from baseline | 18.33 (13.721) | 17.70 (7.589) | 23.75 (21.975)

8. Secondary Outcome: Change in the Fugl-Meyer Motor Total Score (FMMS) Total Score From Baseline at Month 6
Description: The FMMS is used as a clinical measure of body function impairment after stroke that assesses several dimensions of motor impairment, including range of motion in upper and lower limbs, reflex activity, volitional movement, and coordination. The FMMS motor total score ranged from 0 (hemiplegia) to a maximum of 100 points (normal motor performance), and is comprised of a 33-item upper extremity subscale (UE-FMMS) and the 17-item lower extremity subscale (LE-FMMS). Items were scored on a 3-point ordinal scale: 0= cannot perform; 1= partial motion; 2= full motion Individual items are summed to determine scores for the 2 subscale scores, as well as a motor total score (total of the 2 subscales UE-FMMS and LE-FMMS). As a result, the UE-FMMS subscale score ranged from 0 to 66 and the LE-FMMS subscale score ranged from 0 to 34. A maximally affected person will have a score of 0 while a fully functional person will have the highest score (i.e., 34 for LE-FMMS, 66 for UE-FMMS, 100 for FMMS)
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in score on a scale from baseline
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | SB623 Implant (10.0M)
Number analyzed (Participants) | 6 | 6 | 6
Change in score on a scale from baseline | 8.17 (10.834) | 8.67 (4.633) | 17.50 (20.339)

9. Secondary Outcome: Change in the Fugl-Meyer Upper Extremity Motor Function Total Score From Baseline at Month 6
Description: The Fugl-Meyer Upper Extremity subscale (UE-FMMS) is comprised of 33 items that assess several dimensions of motor impairment, including range of motion in upper limbs, reflex activity, volitional movement, and coordination. Scoring is based on direct observation of performance and is scored using a 3-point ordinal scale, where 0=cannot perform; 1=partial motion; and 2=full motion Individual items are summed to provide ranging from 0 (minimum) to 66 (maximum). A maximally affected person will have a score of 0 while a fully functional person will a score of 66.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Change in score on a scale from baseline
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | SB623 Implant (10.0M)
Number analyzed (Participants) | 6 | 6 | 6
Change in score on a scale from baseline | 4.00 (7.321) | 4.50 (3.017) | 11.25 (15.370)

10. Secondary Outcome: Change in the Fugl-Meyer Lower Extremity Motor Function Total Score From Baseline at Month 6
Description: The Fugl-Meyer Lower Extremity subscale (LE-FMMS) is comprised of 17 items that assess several dimensions of motor impairment, including range of motion in lower limbs, reflex activity, volitional movement, and coordination. Scoring is based on direct observation of performance and is scored using a 3-point ordinal scale, where 0=cannot perform; 1=partial motion; and 2=full motion Individual items are summed to provide ranging from 0 (minimum) to 34 (maximum). A maximally affected person will have a score of 0 while a fully functional person will a score of 34.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Change in score on a scale from baseline
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | SB623 Implant (10.0M)
Number analyzed (Participants) | 6 | 6 | 6
Change in score on a scale from baseline | 4.17 (4.355) | 4.17 (3.061) | 6.25 (5.315)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | SB623 Implant (10.0M)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/6 | 2/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SB623 Implant (2.5M) (N=6) | SB623 Implant (5.0M) (N=6) | SB623 Implant (10.0M) (N=6)
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SB623 Implant (2.5M) (N=6) | SB623 Implant (5.0M) (N=6) | SB623 Implant (10.0M) (N=6)
Headache (Nervous system disorders) | 4 | 4 | 3
Muscle spasticity (Nervous system disorders) | 2 | 1 | 1
Convulsion (Nervous system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0
Pneumocephalus (Nervous system disorders) | 0 | 2 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 0
Myoclonus (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Pseudobulbar palsy (Nervous system disorders) | 0 | 1 | 0
Subdural hygroma (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Unresponsive to stimuli (Nervous system disorders) | 0 | 0 | 1
Procedural headache (Injury, poisoning and procedural complications) | 2 | 0 | 3
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 2
Gait disturbance (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Neurological complication associated with device (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Vessel puncture site bruise (General disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 2
Candidiasis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 2 | 1 | 0
C-reactive protein increased (Investigations) | 1 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Lipids increased (Investigations) | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Non-high-density lipoprotein cholesterol increased (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Dissociation (Psychiatric disorders) | 1 | 0 | 0
Emotional distress (Psychiatric disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2014-09-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT01287936/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT01287936/SAP_001.pdf